CLINICAL TRIAL: NCT00838825
Title: Continuous Quality Improvement for Diabetes: Unique Care Delivery Design's Effect on Quality of Care and Utilization of Resources
Brief Title: Continuous Quality Improvement for Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Principal Investigator, Patrick Kearns, Director, Chronic Care Mangement, Santa Clara Valley Health & Hospital System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SCVMC 2/8/08-10
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
Keywords: diabetes; chronic care management; resource utilization; outcome; glycohemoglobin; hospitalization
MeSH Terms: conditions — Diabetes Mellitus | interventions — Case Managers; Chronic Care Model; Delivery of Health Care; Self-Management; Registries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- traditional (No Intervention): The traditional arm is composed of primary care physicians who continue the health care delivery model existing for the 5 years prior to the study. The traditional includes the physician, a pool of resources including random assignment of diabetic educators and includes the entire panel of patients assigned to the PCP.
- care management (Experimental): The care management group is composed of primary care physicians who have been assigned a specific physician extender, the care manager, and an additional medical assistant and form a care manager team working together with registry support, team meetings and instruction in self-management and includes the entire panel of patients assigned to the PCP.
  Interventions: Other: introduction of the chronic care model

INTERVENTIONS:
Other: introduction of the chronic care model — The care management team is organized according to the chronic care model for health care delivery. They are supported by an information registry for diabetes, receive instruction in self-management, have redesigned their work flow to include delegation of functions to care managers who follow specific guidelines and protocols for managing diabetes
  Other Names: care manager; chronic care model; health care delivery; self-management; registry
  Arms: care management

SUMMARY:
The purpose of this study is to compare health care delivery outcomes and costs achieved by two different approaches to health care delivery. The investigators will compare health outcomes for groups of adult patents with diabetes. One group will be managed by our traditional approach to diabetes care. The second group's care delivery is structured according to a design consistent with the Chronic Care Model (CCM).

DETAILED DESCRIPTION:
The study is comparing the effect of an intervention targeting a subset of the diabetic patients within a primary care practice on the resource utilization of resources and disease outcomes on the entire population of patients with diabetes in that practice. The effect will also be compared across the entire panel of patients assigned to the physicians in the 2 arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians practicing in a designated site with > 200 patients assigned to their panel who have been diagnosed with diabetes

Exclusion Criteria:

* Refusal to give informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Primary Completion 2008-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
resource utilization | baseline compared to 2 years intervention

SECONDARY OUTCOMES:
compliance with process measures | 3 years
metabolic outcome | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Kearns, MD, Principal Investigator — Santa Clara Valley Health & Hospital System

IPD SHARING:
Plan to Share IPD: No
Data will be shared in a peer review journal

REFERENCES:
- [Derived] Kearns P. Diabetes Care Management Teams Did Not Reduce Utilization When Compared With Traditional Care: A Randomized Cluster Trial. Manag Care. 2017 Oct;26(10):33-40. PMID 29068297